CLINICAL TRIAL: NCT03884673
Title: Real World Study: Dolutegravir Plus Lamivudine Simplified Therapy in Treatment Experienced HIV-1 Patients
Brief Title: Dolutegravir Plus Lamivudine Simplified Therapy
Status: Recruiting | Type: Observational
Sponsor: Guangzhou 8th People's Hospital (Other)
Collaborators: Shenzhen Third People's Hospital (Other); Dongguan People's Hospital (Other Government); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); The Third People's Hospital of Guilin (Unknown); Guangxi Longtan hospital (Unknown); The Fourth People's Hospital of Nanning (Other); The Third People's Hospital of Kunming (Unknown); Yunnan AIDS Care Center (Other); Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Linghua LI, Vice Chief physician, Guangzhou 8th People's Hospital
Other Study IDs: V2.0-20181215
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: HIV/AIDS
Keywords: DTG + 3TC Simplified Therapy; Simplified Therapy Regimen; Real World Study; HIV-1-infected patients
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DTG+3TC: These cases were given simplified therapy regimen including DTG (50 mg, oral,qd) combined with 3TC (300 mg,oral,qd).
  Interventions: Drug: DTG+ 3TC

INTERVENTIONS:
Drug: DTG+ 3TC — It is a simplified therapy regimen study of dolutegravir combined with lamivudine for HIV-1 infected patients in the real world of China.
  Other Names: A simplified therapy regimen

SUMMARY:
Dolutegravir (DTG) is one type of integrase inhibitor, lamivudine (3TC) is one type of reverse transcriptase inhibitor, both of which are HIV medicine prevents HIV from self-multiplying, reduces the viral load. The data of the existing randomized controlled clinical studies show that the simplified two-drug DTG-based regimen is similar to the three-drug regimen in terms of efficacy, but there are no relevant data and reports on the efficacy and safety of DTG+3TC in HIV-infected patients in China so far. This project aims to explore the efficacy and safety of the DTG + 3TC regimen for HIV-infected patients in real clinical environment, to guide clinical application, and to provide a theoretical basis for the selection of simplified schemes for the formulation of guidelines.

This study was done to see if the combination of two anti-HIV medicines, dolutegravir (DTG, Tivicay) and lamivudine (3TC, Epivir) taken once a day, provide a safe, effective, and well-tolerated treatment for HIV.

DETAILED DESCRIPTION:
This study is an open-label, multicentered, single-arm and phase IV clinical trial. 300 HIV-infected patients who received simplified treatment regimen (50mg DTG+ 400mg 3TC, oral, qd) were selected to observe the treatment efficacy. At week 24, 36, 48 and 96, the rate of viral suppression and CD4 cell count were calculated against baseline. In addition, the safety and drug compliance were also monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Age (> 18 years), male and female;
2. HIV-1 infected;
3. Using a standard three-drug-based regimen for at least 24 weeks. Based on clinical decision making* decide if patients can be treated with the DTG+3TC simplified scheme for a variety of reasons, such as (but not limited to): patients cannot tolerate the conventional three-drug treatment scheme, renal insufficiency, osteoporosis, bone marrow suppression and for other reasons patients cannot use the conventional three-drug treatment scheme;
4. Initial HIV-1 RNA viral load and CD4 cell count were unlimited.
5. CD4 can be monitored at least three times in the first year (including baseline, 24 weeks of treatment and 48 weeks of treatment). After the first year, CD4 can be detected at least once every six months.
6. State Informed Consent for Free Treatment has been signed;
7. Good compliance and signing Informed Consent

(* Reference criteria: Refer to APSIRE study, creatinine clearance rate (> 50 mL/min), no DTG/3TC allergy history, HBsAg negative, no chronic liver disease, no severe liver damage, no pregnancy during the study)

Exclusion Criteria:

1. Has participated in other clinical trials of HIV vaccine or other drug trials in the past three months;
2. Researchers decide if patients could/not complete the scheduled follow-up (factors to consider such as weak, poor compliance, etc.).
3. Has a clear history of DTG or 3TC allergy;
4. HBsAg and/or HBV-DNA positive;
5. Pregnancy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are prescribed to take the simplified therapy regimen (DTG+ 3TC) because they are unable to tolerate the side-effect of or are not fit for the first-line free regimen in China, for example renal failure or osteoporosis, according to clinical judgment, no matter of the HIV-RNA viral loads and CD4 cell counts.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Virus suppression rate | 96 weeks
  ratio of HIV RNA < 50 copies/mL at 48 and 96 weeks of treatment
Adverse events | 96 weeks
  Rate of adverse events reported during the observational period

SECONDARY OUTCOMES:
The immunological ability (CD4+) | 96 weeks
  CD4 cell count (baseline to 48 weeks and 96 weeks)
Drug compliance | 96 weeks
  To explicit the number of people who have completed the treatment
The immunological ability (CD8+) | 96 weeks
  CD4 +/ CD8 + ratio (baseline to 48 weeks and 96 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Cai, Bachelor, Principal Investigator — Guangzhou 8th People's Hospital
Locations (1):
- Guangzhou 8th People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cahn P, Madero JS, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man C, Currie A, Underwood M, Tenorio AR, Pappa K, Wynne B, Fettiplace A, Gartland M, Aboud M, Smith K; GEMINI Study Team. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferiority, phase 3 trials. Lancet. 2019 Jan 12;393(10167):143-155. doi: 10.1016/S0140-6736(18)32462-0. Epub 2018 Nov 9. PMID 30420123
- [Background] Cahn P, Rolon MJ, Figueroa MI, Gun A, Patterson P, Sued O. Dolutegravir-lamivudine as initial therapy in HIV-1 infected, ARV-naive patients, 48-week results of the PADDLE (Pilot Antiretroviral Design with Dolutegravir LamivudinE) study. J Int AIDS Soc. 2017 May 9;20(1):21678. doi: 10.7448/IAS.20.01.21678. PMID 28537061
- [Background] Taiwo BO, Zheng L, Stefanescu A, Nyaku A, Bezins B, Wallis CL, Godfrey C, Sax PE, Acosta E, Haas D, Smith KY, Sha B, Van Dam C, Gulick RM. ACTG A5353: A Pilot Study of Dolutegravir Plus Lamivudine for Initial Treatment of Human Immunodeficiency Virus-1 (HIV-1)-infected Participants With HIV-1 RNA <500000 Copies/mL. Clin Infect Dis. 2018 May 17;66(11):1689-1697. doi: 10.1093/cid/cix1083. PMID 29253097